CLINICAL TRIAL: NCT00351039
Title: Phase I/II Trial of Bevacizumab, Pemetrexed and Erlotinib in the First-Line Treatment of Elderly Patients With Advanced (Stage IIIB(With Malignant Pleural Effusion) or IV) Non-Squamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Phase I/II Trial of Bevacizumab, Pemetrexed and Erlotinib in Elderly Patients With Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Genentech, Inc. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14659
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Results first posted 2010-08-30 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2010-08

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Erlotinib Hydrochloride; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab, Erlotinib, Pemetrexed (Experimental): Single Arm Phase II trial in elderly patients with advanced stage Non-Squamous Non-Small Cell Lung Cancer
  Interventions: Drug: Bevacizumab; Drug: Erlotinib; Drug: Pemetrexed

INTERVENTIONS:
Drug: Bevacizumab — Treatment Regimen Item 1: Bevacizumab 10 mg/Kg I. V. Day 1 and Day 15. Repeat cycles every 28 days.
  Other Names: Avastin
Drug: Erlotinib — Treatment Regimen Item 2: Erlotinib 150mg Per Orally (PO) Once Daily (QD) for 7 days starting day 2 and day 15. Repeat cycles every 28 days.
  Other Names: Tarceva
Drug: Pemetrexed — Treatment Regimen Item 3: Premetrexed 500mg/m2 I.V. Day 1 and Day 15. Repeat cycles every 28 days.
  Other Names: Alimta

SUMMARY:
This is a Phase I/II trial of elderly patients (> 70 years of age). Patients in this age group with previously un-treated Advanced Stage Non-Squamous Non-Small Cell Lung Cancer (NSCLC) with Stage IIIB (with malignant pleural effusion) and stage IV disease will be enrolled. Therapy consists of three drugs (Premetrexed[Alimta™], Bevacizumab and Erlotinib[Tarceva™]) which are given every 28 days.

DETAILED DESCRIPTION:
This is a Phase I/II trial of elderly patients (> 70 years of age) with previously un-treated Advanced Stage Non-Squamous NSCLC with Stage IIIB (with malignant pleural effusion) and stage IV disease will be enrolled.

Treatment Regimen:

Premetrexed (Alimta™) 500 milligrams(mg)/Meter squared(m20 Intravenous(I.V.) Day 1 and Day 15; Bevacizumab 10mg/Kilogram(Kg) I. V. Day 1 and Day 15; Erlotinib (Tarceva™) 150mg Per Orally(PO) Once Daily(QD) for 7 days starting day 2 and day 15; Repeat cycles every 28 days.

All three drugs will be continued for two cycles after maximal response. After which patient will be maintained only on the Bevacizumab and Erlotinib until progression. If patient has stable disease after the first two cycles then patient will be given another two cycles with all three drugs before maintenance treatment with Bevacizumab and Erlotinib is initiated.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically proven diagnosis of Non-Squamous NSCLC. NSCLC histologies that will be included in this trial will be adenocarcinoma, large cell carcinoma and adeno-squamous carcinoma. Patients with bronchioloalveolar carcinoma (BAC) will be also included in this trial.
* Patients must be 70 years of age or older.
* Patient must have either stage IIIB disease with malignant pleural effusion or stage IV disease. All patients must have measurable disease. Evaluable disease will be separately outlined and elucidated.
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of either 0 or 1.
* Patient must have adequate renal function with a serum creatinine level of less than 1.5mg/dl and patient should have a calculated creatinine clearance of more than 45ml/min.
* Patient must have adequate hepatic function with a serum bilirubin level of less that 3mg/dl, and an alkaline phosphatase, Alanine Amino Transferase (ALT) and Aspartate Amino Transferase (AST) of less than three times the upper limit of normal
* Patient must also have evidence of adequate bone marrow function with an absolute neutrophil count of more than 1, 500 cells per deciliter and a platelet count of more than 100,000 per deciliter.
* Patients must be more than 28 days since prior open biopsy; more than 7 days since prior fine-needle aspiration; more than 7 days since prior core biopsy; more than 28 days since prior surgery.
* Patients must be able to take dexamethasone, folic acid and vitamin B-12 supplementation.
* All patients must sign informed consent that will detail the investigational nature of the study in accordance with the institutional and federal guidelines.

Exclusion Criteria:

* Lung carcinoma of squamous cell histology or any histology in close proximity to a major vessel, with or without cavitation.
* Patients with hypercalcemia (corrected calcium of more than 11 mg/dl) will be excluded.
* Patients with history of hemoptysis, hematemesis, coagulopathy or thrombosis will be excluded.
* Patients requiring anticoagulation for any reason will be excluded.
* Patients who recently have an acute infection.
* History of palliative radiation therapy within 2 weeks.
* Blood pressure of >150/100 Millimeter Mercury(mmHg).
* Currently ongoing unstable angina.
* New York Heart Association (NYHA) Grade II or greater congestive heart failure.
* History of myocardial infarction within 6 months.
* History of stroke within 6 months.
* Clinically significant peripheral vascular disease.
* Presence of central nervous system or brain metastases.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study.
* Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to Day 0.
* Pregnant (positive pregnancy test) or lactating.
* Urine calculated creatinine clearance of less than 45ml/minute and a urinary protein. Creatinine ratio of more than 1.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 1.
* Serious, non-healing wound, ulcer, or bone fracture.
* Inability to comply with study and/or follow-up procedures.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Simon, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffiitt Cancer Center Clinical Trials Website — http://www.moffitt.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: July 2006 through September 2008 at Moffitt Cancer Center
Pre-assignment Details: Phase I run-in. One participant was excluded due to screen failure, showing that they should not have been included to start.
Groups:
- Experimental: Bevacizumab, Erlotinib, Pemetrexed: Treatment Regimen Item 1: Bevacizumab 10mg/Kg I. V. Day 1 and Day 15. Repeat cycles every 28 days. Treatment Regimen Item 2: Erlotinib(Tarceva™) 150mg Per Orally (PO) Once Daily (QD) for 7 days starting day 2 and day 15. Repeat cycles every 28 days. Treatment Regimen Item 3: Pemetrexed(Alimta™) 500mg/m2 I.V. Day 1 and Day 15. Repeat cycles every 28 days. The regimen then was modified to the following dose:
  Bevacizumab 15mg/kg Day 1 every 21 days (Q21); Pemetrexed 500 mg/m2 Day 1 Q 21; Erlotinib 150 mg QD PO Day 2 to day 15 (Both days inclusive). This dose was then recommended to be Phase II dose.
Period: Overall Study
Arm/Group | Experimental: Bevacizumab, Erlotinib, Pemetrexed
Started | 8
Completed | 8 (The study was halted before Phase II was initiated.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: Bevacizumab, Erlotinib, Pemetrexed
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 75 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 8
Number of Participants who received treatment on this protocol [Number; unit: Participants] — All patients accrued sought and received treatment at the Moffitt Cancer Center.
  Participants | 8

OUTCOME MEASURES:

1. Secondary Outcome: One-year Survival(1-year S)
Description: Secondary Objective: One-year survival(1-year S) in patients with advanced NSCLC treated with this regimen.
Time Frame: 26 Months
Population: Had the study been completed as planned we would have measured the One-year Survival. This study was closed early due to poor accrual.
Groups:
- Experimental: Bevacizumab, Erlotinib, Pemetrexed: Treatment Regimen Item 1: Bevacizumab 10mg/Kg I. V. Day 1 and Day 15. Repeat cycles every 28 days. Treatment Regimen Item 2: Erlotinib(Tarceva™) 150mg PO QD for 7 days starting day 2 and day 15. Repeat cycles every 28 days. Treatment Regimen Item 3: Pemetrexed(Alimta™) 500mg/m2 I.V. Day 1 and Day 15. Repeat cycles every 28 days. The regimen then was modified to the following dose:
  Bevacizumab 15mg/kg Day 1 Q21 Pemetrexed 500 mg/m2 Day 1 Q 21 Erlotinib 150 mg QD PO Day 2 to day 15 (Both days inclusive) This dose was then recommended to be phase II dose.
Arm/Group | Experimental: Bevacizumab, Erlotinib, Pemetrexed
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Patients Who Responded to Treatment
Description: Phase I:
  Response Evaluation Criteria In Solid Tumors (RECIST)Criteria was used for Response. Partial Response (PR) is defined as at least a 30% decrease in the sum of Longest Dimention (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: 26 Months
Population: 8 patients were accrued to the Phase I component of the trial. No patients were accrued to the Phase II component of the trial.
Arm/Group | Experimental: Bevacizumab, Erlotinib, Pemetrexed
Number analyzed (Participants) | 0

3. Secondary Outcome: Quality of Life (QOL)
Description: The Scales we were intending to use were:
  Instrumental Activities of Daily Living (IADL): Range of Scale 0 (Best) to 8 (Worst).
  Cumulative Illness Rating Scale-Geriatric (CIRS-G): Range of Scores 1(Best) to 18 (Worst).
  Functional Assessment of Cancer Therapy-Lung (FACT-L): Range of Scores 0 (Best) to 48 (Worst).
  Fatigue Symptom Inventory (FSI): Range of Scores 0(Best) to 121 (Worst).
  Each scale would have been evaluated independently. Since the study was not completed and closed early due to poor accrual, none of the QOL parameters were analyzed.
Time Frame: 26 Months
Population: Since no patients were accrued to the Phase II component of the trial, 0 patients were analyzed for these scales.
Arm/Group | Experimental: Bevacizumab, Erlotinib, Pemetrexed
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Grade 3 and Grade 4 Adverse Events
Description: By Safety, the intent was to capture, tabulate, list all of the grade 3 and 4 adverse effects seen by this protocol. For each toxicity, we followed the Common Toxicity Criteria(NCI CTC)Version 2.0 Toxicity scale guidelines.
Time Frame: 26 Months
Population: This study was initially intended to be a Phase I/II study with a brief Phase I Run-in. After the brief Phase I Run-in the study was closed without initiating the Phase II component.
Measure: Number; unit: Participants
Arm/Group | Experimental: Bevacizumab, Erlotinib, Pemetrexed
Number analyzed (Participants) | 8
Participants | 8

5. Primary Outcome: Progression Free Survival (PFS)
Description: The primary objective was to determine the progression free survival (PFS), in newly diagnosed patients with advanced Non Small Cell Lung Cancer (NSCLC) who are treated with a regimen consisting of Bevacizumab(B), pemetrexed(A), and erlotnib(T). This was a Phase I/II study. This trial was halted after the Phase I component was completed. The Phase II component was never initiated.
Time Frame: 26 months
Population: No patients proceeded to Phase II for evaluation.
Arm/Group | Experimental: Bevacizumab, Erlotinib, Pemetrexed
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival (Median Survival [MS])
Description: Secondary Objective: Determine the Overall Survival (median survival[MS]) in patients with advanced NSCLC treated with this regimen. Patients were to be followed until death and survival curves were to be generated.
Time Frame: 26 Months
Population: Had the study been completed as planned we would have measured Overall Survival described as Median Survival. This study was closed early due to poor accrual.
Arm/Group | Experimental: Bevacizumab, Erlotinib, Pemetrexed
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 26 months
Description: All noted adverse events were reported on the accrued patients. Hence the threshold is Zero.
Arm/Group | Experimental: Bevacizumab, Erlotinib, Pemetrexed
Serious Adverse Events (participants affected / at risk) | 6/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Bevacizumab, Erlotinib, Pemetrexed (N=8)
Syncope (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Unlikely
Non Febrile Neutropenia (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Causality: Definitely Related
Fatigue (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Causality: 2 Definitely Related, 1 Probably Related
Dyspnea with exertion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Definitely Related
Proteinuria (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Probably Related
Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Possibly Related
Hyperglycemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Unrelated
Pain, Penis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Unrelated
Secondary Malignancy (bladder tumor) (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Unrelated
Right Hip Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Unrelated
Dehydration (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Probably Related
Anorexia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Probably Related
Hypokalemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Probably Related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Bevacizumab, Erlotinib, Pemetrexed (N=8)
Pruritis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Probably Related
Fatigue (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Causality: 1 Definitely Related, 1 Probably Related, 1 Unrelated
Mucositis (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Causality: 1 Probably Related, 1 Possibly Related
Anemia (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Causality: 1 Definitely Related, 1 Unlikely
Generalized Weakness (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Definitely Related
Nausea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Probably Related
Vomiting (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Probably Related
Expressive Aphasia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Unlikely
Neutropenia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Probably Related
Serum Creatinine Elevation (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Probably Related
ALT Elevation (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Probably Related
Non Febrile Neutropenia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Probably Related
Bilateral Lower Extremity Weakness (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Unlikely
Proteinuria (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Probably Related
Hyperglycemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Unrelated
Pain, Left Axillary Area (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Unrelated
Pain, Back (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Unrelated
Constipation (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Unrelated
Left Hip Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Unrelated
Gingival Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Unrelated
Hypernatremia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality:Probably Related
Rash-Acneiform (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Definitely Related
Yeast Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Unrelated

LIMITATIONS AND CAVEATS:
This study was closed early due to poor accrual. The recommended Phase II dose was determined after the brief Phase I run-in, but the Phase II component of this study was never initiated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No